CLINICAL TRIAL: NCT00328731
Title: The Effectiveness of Milk Allergy Elimination Through NAET Treatments
Brief Title: Milk ALLERGY ELIMINATION THROUGH NAET® (Nambudripad's Allergy Elimination Techniques).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nambudripad's Allergy Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAR Foundation study 120
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2006-05-22 (Estimated); Status verified 2005-01

CONDITIONS: Milk Allergy
Keywords: Allergy; NAET
MeSH Terms: conditions — Milk Hypersensitivity; Hypersensitivity | interventions — Methods

INTERVENTIONS:
Procedure: Procedure

SUMMARY:
We sought to determine the efficacy of NAET® in permanently eliminating milk allergy for a sample of patients.

We hypothesize that the subjects in the experimental group will show similar level of allergies and sensitivities initially on all nine diagnostic measures used here. After receiving the NAET treatments, the Experimental group will demonstrate a significant reduction in the milk sensitivities and allergies when compared to the control group at the final evaluation using same diagnostic measures.

DETAILED DESCRIPTION:
Background: Although several standard clinical techniques are used to detect and treat common allergic conditions, each one is limited in scope and requires to follow repeated treatment protocols. The non-invasive system known as NAET® does not generally have such limitations and has over the last twenty-three years been demonstrated to be effective clinically in thousands of cases. NAET® is a natural treatment that utilizes standard medical diagnostic measures along with kinesiolgocal, chiropractic and oriental testing, procedures to identify the allergens, as well as the intensity of reactions to the allergens which vary from individual to individual. Treatment consists of a sequence of spinal manipulations at specific thoracic and lumbar spinal levels along with acupuncture acupressure on configurations of standard acupuncture points.

Methods: In a double blind study, 26 patients with diagnosed milk allergy (13 males, 13 females, age range between 18-65 years) were randomly assigned to 2 groups:

1. NAET®/Experimental group, and
2. Placebo/control group The study was conducted by 12 volunteer-clinicians from NAET Research associates, divided into six investigator groups. Each group conducted a designated sequential part of the study independently from all other groups, that is, was blinded from all other groups for the duration of the study. Subjects from both groups (Experimental and Control) were evaluated immediatedly before treatment and eight weeks thereafter using the following nine diagnostic measures: Subjective history (Allergy Symptom Rating Scale or ASRS); ALCAT Test; antibodies to milk protein in the blood serum by Immunoglobulins G, Immunoglobulins A, Immuno-globulins M, and Immunoglobulins E (IgG, IgA, IgM, IgE) by Elisa method (enzyme linked Immunozorbant Assay); Intradermal testing for milk sensitivity. NSTRS (Kinesiological muscle response testing also known as Neuromuscular Sensitivity Testing) and Pulse difference Rating Scale (PDRS) were tested by two well trained NST clinicians at two different times before and after the treatments. Both groups demonstrated allergic sensitivities to whole milk test sample in varying degrees. After completing the evaluations, the Experimental group received 2 NAET® treatments on whole milk, on two consecutive Saturdays. The Placebo group received two treatments on placebo samples on the same days along with the experimental group on two consecutive Saturdays as well. At the end of the treatment phase, once again both groups were evaluated for whole milk test sample using all of the nine diagnostic measures.

Results On the nine diagnostic measures there was a significant difference in the means of the before and after measures of the Experimental group, while they remained almost the same for the Placebo group. At 95% CI, p-values were less than 0.05 in all tests except for IgG study (p-value=1.30). NSTRS and PDRS were evaluated by two clinicians at different time to evaluate the intertester relability among two clinicians for these two tests. A significant correlation was noticed with the results both testers received on these two testing-NST and PDRS (p-value <0.0001).

Conclusion The study demonstrated the efficacy of eliminating or reducing milk allergy using the NAET® treatment protocol. This study also evaluated the reliability of performing two testing procedures (NST & PDRS) by two independent examiners in testing the subjects for milk at two different times. There was a significant correlation in the results they received as shown above, when the two clinicians tested the subjects independently, demonstrating that there is a good reliability between these well trained clinicians in their performance while doing these two evaluations.

ELIGIBILITY:
Inclusion Criteria:

Known milk allergy, sensitivity or intolerances. -

Exclusion Criteria:

No milk allergy or sensitivity H/o Anaphylaxis or severe reactions Any other major illnesses preventing from taking part in any study

-

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26
Dates: Start 2005-01; Study Completion 2006-01

PRIMARY OUTCOMES:
Reduction of Milk allergies

SECONDARY OUTCOMES:
This study also evaluated the reliability of performing two testing procedures (NST & PDRS) by two independent examiners in testing the subjects for milk at two different times.

CONTACTS AND LOCATIONS:
Overall Officials: Devi S Nambudripad, DC,PhD,L.Ac, Principal Investigator — NAR Foundation
Locations (1):
- NAET-Pain Clinic, Buena Park, California, United States